CLINICAL TRIAL: NCT04042740
Title: Glecaprevir/Pibrentasvir Fixed-dose Combination Treatment for Acute Hepatitis C Virus Infection (PURGE-C)
Brief Title: Glecaprevir/Pibrentasvir Fixed-dose Combination Treatment for Acute Hepatitis C Virus Infection
Acronym: PURGE-C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: AbbVie (Industry); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5380; 38553 (Registry Identifier: DAIDS-ES Registry Number); UM1AI068636 (NIH)
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Results first posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Hepatitis C Infection; HIV Infection
Keywords: Acute Hepatitis C Infection; Glecaprevir; Pibrentasvir; 4 weeks; Direct-acting antivirals
MeSH Terms: conditions — Hepatitis C; HIV Infections | interventions — glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Glecaprevir/Pibrentasvir (G/P) (Experimental): Participants were assigned to receive G/P FDC tablets to be taken orally once daily for 4 weeks (Step 1).
  Participants who experienced HCV re-infection, suspected relapse, virologic failure, or undefined post-treatment viremia in Step 1 were offered to enter Step 2 for re-treatment. HCV re-treatment regimens may have included G/P FDC tablets orally once daily for 8-16 weeks, or alternate regimens through clinical care.
  Interventions: Drug: Glecaprevir/Pibrentasvir (G/P)

INTERVENTIONS:
Drug: Glecaprevir/Pibrentasvir (G/P) — Fixed-dose combination (FDC) tablets containing 100 mg of glecaprevir and 40 mg of pibrentasvir; administered as 3 tablets orally.
  Other Names: Mavyret

SUMMARY:
The purpose of this study was to assess the efficacy of a fixed dose combination (FDC) of glecaprevir/pibrentasvir (G/P) given for 4 weeks for treatment of acute hepatitis C (HCV), with or without HIV-1 coinfection.

DETAILED DESCRIPTION:
The study was conducted in two steps. In Step 1, participants received four weeks of treatment with G/P for acute HCV infection and were then followed 24 weeks post treatment. Participants with HCV recurrence (reinfection, suspected relapse or undefined post-treatment viremia) or HCV virologic failure before or at the Step 1 Week 16 entered Step 2 and were offered HCV re-treatment. The remaining participants were followed in Step 1 for a total of 28 weeks. The study primary and secondary outcome measures pertain to Step 1.

In Step 2, participants were re-treated for up to 16 weeks (G/P or alternate regimen through standard of care), and were followed for 24 weeks post treatment. This post-treatment follow-up included a visit for the determination of HCV sustained virologic response (SVR12) after re-treatment. All summaries of data captured from Step 2 are pooled across HCV re-treatment regimens, as specified in the Statistical Analysis Plan.

In Step 1, study visits were scheduled at study entry, weeks 1 and 2 (on-treatment), week 4 (treatment discontinuation), and weeks 8, 12, 16 and 28 (post-treatment follow-up). In Step 2, participants had study visits during the re-treatment period, where the number of visits depended on the re-treatment regimen, and at weeks 12 and 24 post treatment. Study visits included physical examinations, clinical assessments, blood and urine collection, questionnaires, and HCV re-infection prevention counseling.

ELIGIBILITY:
Inclusion Criteria

* Acute HCV infection (or reinfection) within 24 weeks prior to entry
* Detectable HCV RNA at the screening visit

Exclusion Criteria

* Any HCV treatment during the current acute HCV infection episode
* Known preexisting cirrhosis
* Acute HIV-1 infection
* Presence of active or acute AIDS-defining opportunistic infections, active serious infection (other than HIV-1 or HCV), active hepatitis B virus (HBV) or active hepatitis A virus (HAV)
* Chronic use of systemically administered immunosuppressive agents
* History of solid organ transplantation
* History of conditions that could interfere with the absorption of the study drug
* Concurrent use of prohibited medications
* Known hypersensitivity to glecaprevir or pibrentasvir, the metabolites, or parts of the formulation
* Females who are pregnant or breastfeeding
* Males with pregnant female partner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Y. Kim, MD, Study Chair — Massachusetts General Hospital (MGH) CRS; Susanna Naggie, MD, MHS, Study Chair — Duke University Medical Center CRS; David Wyles, MD, Study Chair — University of Colorado Hospital CRS
Locations (12):
- United States (11):
  - Ucsd, Avrc Crs (701), San Diego, California
  - University of California, San Francisco HIV/AIDS CRS (801), San Francisco, California
  - University of Colorado Hospital CRS (6101), Aurora, Colorado
  - Whitman-Walker Institute, Inc. CRS (31791), Washington D.C., District of Columbia
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS (101), Boston, Massachusetts
  - Weill Cornell Chelsea CRS (7804), New York, New York
  - Columbia Physicians and Surgeons CRS (30329), New York, New York
  - Weill Cornell Upton CRS (7803), New York, New York
  - Unc Aids Crs (3201), Chapel Hill, North Carolina
  - University of Washington AIDS CRS (1401), Seattle, Washington
- Instituto de Pesquisa Clinica Evandro Chagas (12101), Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and throughout period of funding of the ACTG Network by NIH.
Access Criteria: * With whom?
    * Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses?
    * To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available?
    * Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://actgnetwork.org/about-actg/templates-and-forms. Researchers of approved proposals will need to sign an ACTG Data Use Agreement before receiving the data.

REFERENCES:
- [Derived] Kim AY, Kang M, Umbleja T, Nunes EP, Marks KM, Luetkemeyer AF, Koebele C, Wimbish C, Fierer DS, Kliemann DA, Solomon SS, Kort J, Kiser JJ, Lauer GM, Chung RT, Sowah LA, Alston-Smith BL, Wyles DL, Naggie S; A5380 Study Team. Short Course Therapy With Glecaprevir/Pibrentasvir for Early Hepatitis C Virus Infection: PURGE-C. Clin Infect Dis. 2025 Jul 30:ciaf305. doi: 10.1093/cid/ciaf305. Online ahead of print. PMID 40736252
- See also: Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017 — https://rsc.niaid.nih.gov/sites/default/files/daids-ae-grading-table-v2-nov2014.pdf
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — https://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from November 2019 to January 2023.
Groups:
- Glecaprevir/Pibrentasvir (G/P) Followed by Re-treatment, as Needed: G/P FDC tablets to be taken orally once daily for 4 weeks, followed by 24 weeks of observation (Step 1).
  Participants who experienced HCV re-infection, suspected relapse, virologic failure, or undefined post-treatment viremia were offered re-treatment (8-16 weeks), followed by 24 weeks of observation (Step 2).
Period: Step 1 (4-week G/P + 24-week Follow-up)
Arm/Group | Glecaprevir/Pibrentasvir (G/P) Followed by Re-treatment, as Needed
Started | 45
Initiated Study Treatment | 45
Completed 16 Weeks | 44
Completed | 42
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1
Period: Step 2 (HCV Re-treatment)
Arm/Group | Glecaprevir/Pibrentasvir (G/P) Followed by Re-treatment, as Needed
Started | 4 (Participants with HCV re-infection, suspected relapse, virologic failure, or undefined post-treatment viremia in Step 1 were offered re-treatment in Step 2.)
Completed | 3
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: All eligible participants who initiated study treatment
Groups:
- Glecaprevir/Pibrentasvir (G/P): G/P FDC tablets to be taken orally once daily for 4 weeks, followed by 24 weeks of observation (Step 1).
Arm/Group | Glecaprevir/Pibrentasvir (G/P)
Number analyzed (Participants) | 45
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Age at study enrollment
  years | 36 [29 to 43]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender identity by participant self-report
  Participants
    Female | 1
    Male | 43
    Non-binary | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Sex assigned at birth
  Participants
    Female | 1
    Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race (US NIH/OMB definition), expanded for non-US regions
  Participants
    Asian | 3
    Black or African American | 12
    White | 23
    Other | 4
    Unknown | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31
  Brazil | 14
HCV history [Count of Participants; unit: Participants]
  No history of HCV | 38
  Previous HCV | 7
HCV genotype [Count of Participants; unit: Participants]
  Genotype 1 | 32
  Genotype 2 | 2
  Genotype 3 | 1
  Genotype 4 | 5
  Indeterminate | 1
  Not detected | 3
  Unable to result | 1
HCV RNA [Median (Inter-Quartile Range); unit: log10 IU/mL] | 5.25 [3.30 to 6.00]
HIV-1 status [Count of Participants; unit: Participants]
  HIV-1 present | 23
  No HIV-1 | 22
Injection drug use [Count of Participants; unit: Participants]
  Former | 12
  Never | 33

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response at 12 Weeks Post Treatment Discontinuation (SVR12)
Description: SVR12 defined as unquantifiable HCV RNA (less than the lower limit of quantification [LLOQ], target detected [TD] or target not detected [TND]) at study visit 12 weeks post treatment (Week 16). If a participant did not have HCV RNA measurement at Week 16, the participant was considered as SVR12 failure, unless there were preceding and subsequent HCV RNA measurements that were both LLOQ (either TD or TND).
Time Frame: Week 16 (12 weeks post study treatment)
Population: All eligible participants who initiated study treatment
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir/Pibrentasvir (G/P)
Number analyzed (Participants) | 45
percentage of participants | 84.4 [73.6 to 91.3]

2. Primary Outcome: Percentage of Participants Who Experienced Adverse Events (AEs)
Description: Study protocol required reporting of (1) AEs Grade greater than or equal to 2, (2) AEs that led to a change in study treatment regardless of grade and (3) AEs meeting ICH definition of serious AE (SAE) or Expedited AE (EAE) reporting requirement. DAIDS AE Grading Table (V2.1) and DAIDS EAE Manual (V2.0) were used.
Time Frame: From study entry to Week 8 (4 weeks post study treatment)
Population: All eligible participants who initiated study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir/Pibrentasvir (G/P)
Number analyzed (Participants) | 45
percentage of participants | 60.0 [45.5 to 73.0]

3. Primary Outcome: Number of Participants Who Completed 4 Weeks of Treatment Without Discontinuation Due to AEs
Description: Number of participants who completed 4 weeks of treatment without discontinuation due to AEs
Time Frame: From study entry to Week 4
Population: All eligible participants who initiated study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Glecaprevir/Pibrentasvir (G/P)
Number analyzed (Participants) | 45
Participants | 45

4. Secondary Outcome: Percentage of Participants With HCV RNA Less Than LLOQ
Description: Percentage of participants with HCV RNA less than LLOQ (TD or TND). Given the substantial amount of missing data due to the SARS-CoV-2 pandemic, the planned analysis of 90% confidence intervals for the percentage of participants with HCV RNA <LLOQ at study visits could not be conducted in a meaningful way.
Time Frame: Weeks 1, 2, 4, 8, 12, 28
Population: All eligible participants who initiated study treatment with HCV RNA data available at the given visit. The study conduct overlapped with the COVID-19 pandemic. At the beginning of the COVID-19 pandemic, Week 16 visit was prioritized; other study visits may have occurred remotely without HCV RNA collection, due to COVID-related restrictions at the sites.
Measure: Number; unit: percentage of participants
Arm/Group | Glecaprevir/Pibrentasvir (G/P)
Number analyzed (Participants) | 45
percentage of participants
  Week 1 HCV RNA <LLOQ: number analyzed (Participants) | 37
  Week 1 HCV RNA <LLOQ | 51.4
  Week 2 HCV RNA <LLOQ: number analyzed (Participants) | 41
  Week 2 HCV RNA <LLOQ | 70.7
  Week 4 HCV RNA <LLOQ: number analyzed (Participants) | 41
  Week 4 HCV RNA <LLOQ | 97.6
  Week 8 HCV RNA <LLOQ: number analyzed (Participants) | 36
  Week 8 HCV RNA <LLOQ | 97.2
  Week 12 HCV RNA <LLOQ: number analyzed (Participants) | 34
  Week 12 HCV RNA <LLOQ | 88.2
  Week 28 HCV RNA <LLOQ: number analyzed (Participants) | 42
  Week 28 HCV RNA <LLOQ | 81.0

5. Secondary Outcome: Number of Participants With HCV Virologic Failure
Description: Virologic failure defined as failure to achieve unquantifiable HCV RNA or confirmed increase in HCV RNA greater than 1 log10 from on-treatment nadir
Time Frame: From Week 1 to Week 16
Population: All eligible participants who initiated study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Glecaprevir/Pibrentasvir (G/P)
Number analyzed (Participants) | 45
Participants | 6

6. Other Pre Specified Outcome: Number of Participants by HCV Re-Treatment Regimen in Step 2
Description: Participants who experienced HCV re-infection, suspected relapse, virologic failure, or undefined post-treatment viremia in Step 1 were offered to enter Step 2 for re-treatment. HCV re-treatment regimens may have included various regimens including study-provided G/P and alternate regimens through clinical care. This outcome measure is used to report the re-treatment regimens observed in Step 2.
Time Frame: At Step 2 entry (median time of Step 2 entry was at 21 weeks after study entry.
Population: All participants who entered Step 2 for HCV re-treatment.
Measure: Count of Participants; unit: Participants
Groups:
- HCV Re-Treatment Regimens: Participants who experienced HCV re-infection, suspected relapse, virologic failure, or undefined post-treatment viremia in Step 1 were offered to enter Step 2 for re-treatment. HCV re-treatment regimens may have included G/P FDC tablets orally once daily for 8-16 weeks, or alternate regimens through clinical care.
Arm/Group | HCV Re-Treatment Regimens
Number analyzed (Participants) | 4
Participants
  Glecaprevir/pibrentasvir | 3
  Sofosbuvir/velpatasvir/voxilaprevir | 1

ADVERSE EVENTS:
Time Frame: Step 1: From study entry to study completion or Step 2 entry or premature study discontinuation (median time in Step 1 was 28 weeks). Step 2: From Step 2 entry to study completion or premature discontinuation (median time in Step 2 was 21 weeks).
Description: New diagnoses, signs/symptoms and laboratory values that were Grade ≥2, led to a change in study treatment regardless of grade or met SAE definition or EAE reporting requirements, regardless of attribution to study treatment. DAIDS AE Grading Table (V2.1) and EAE Manual (V1.0) were used. All eligible participants who initiated study treatment are included. For the subset who continued to Step 2 for HCV re-treatment, the AEs that occurred in Step 2 are shown in a separate column.
Arm/Group | Glecaprevir/Pibrentasvir (G/P) | HCV Re-Treatment Regimens
All-Cause Mortality (participants affected / at risk) | 0/45 | 4/4
Serious Adverse Events (participants affected / at risk) | 4/45 | 1/4
Other Adverse Events (participants affected / at risk) | 32/45 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Glecaprevir/Pibrentasvir (G/P) (N=45) | HCV Re-Treatment Regimens (N=4)
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Carotid artery disease (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Glecaprevir/Pibrentasvir (G/P) (N=45) | HCV Re-Treatment Regimens (N=4)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 1
Proctitis (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Anal chlamydia infection (Infections and infestations) | 1 | 0
Anal gonococcal infection (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 5 | 0
Cellulitis (Infections and infestations) | 0 | 1
Gonorrhoea (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Monkeypox (Infections and infestations) | 2 | 0
Orchitis (Infections and infestations) | 1 | 0
Oropharyngeal gonococcal infection (Infections and infestations) | 1 | 1
Otitis externa (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Proctitis chlamydial (Infections and infestations) | 1 | 0
Proctitis gonococcal (Infections and infestations) | 1 | 1
Proctitis herpes (Infections and infestations) | 0 | 1
Purulent discharge (Infections and infestations) | 1 | 0
Rash pustular (Infections and infestations) | 1 | 0
Secondary syphilis (Infections and infestations) | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urethritis chlamydial (Infections and infestations) | 1 | 0
Urethritis gonococcal (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 2 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 9 | 1
Aspartate aminotransferase increased (Investigations) | 6 | 0
Bilirubin conjugated increased (Investigations) | 3 | 0
Blood bilirubin increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 2 | 0
Blood sodium decreased (Investigations) | 1 | 0
Creatinine renal clearance (Investigations) | 1 | 0
Creatinine renal clearance decreased (Investigations) | 8 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Lipase increased (Investigations) | 2 | 0
Prothrombin time prolonged (Investigations) | 1 | 0
Weight increased (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Inguinal mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 1
Glycosuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Genital pain (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0
Penile ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
High risk sexual behaviour (Social circumstances) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT04042740/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT04042740/SAP_001.pdf